CLINICAL TRIAL: NCT05495659
Title: Clinical Study of GREE(a Name of Chinese Company)-AI(Artificial Intelligence) Medical Software in the Detection of Ureteral Stent Encrustation
Brief Title: Detection of Ureteral Stent Encrustation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Minbo Yan, Clinical Professor, Fifth Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: FSYS-2022-K122-1
Record Dates: First submitted 2022-07-31; First posted 2022-08-10 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Ureteral Stent-Related Symptom
Keywords: GREE-AI medical software, ureteral stent, encrustation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Ureteral stents are the most commonly used postoperative implantable materials in urology. The indwelling ureteral stents often lead to the formation of encrustation, with an incidence of 10%, which will lead to complications such as obstruction, lower urinary tract symptom (LUTS）, and difficulty in extubation. At present, there is no accurate and sensitive diagnostic criteria for ureteral stents encrustation. Previously, we developed the artificial intelligence-based ureteral stents encrustation identification software - GREE-AI Medical Software (GAIMS) with the collaboration of GREE ELECTRIC APPLIANCES,INCORPORATED.OF ZHUHAI(a city of Guangdong, China). In order to further evaluate the diagnostic sensitivity and accuracy of the software in practical clinical applications, and to verify its predictive ability for ureteral stents encrustation, the following single-center, prospective, double-blind, diagnostic cohort study is planned.

This study will use the gold standard as a reference to evaluate the sensitivity and specificity of GAIMS for detecting ureteral stents encrustation. At the same time, it will be compared with non-enhanced contrast Computed Tomography examinations interpreted by clinical radiologists to evaluate the pros and cons of GAIMS in detecting ureteral stents encrustation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who plan to undergo ureteral stent placement due to urinary calculi or urinary system obstruction;
2. Aged over 12 years old;
3. The estimated time of ureteral stent placement is more than 2 weeks but less than 1 year;
4. Voluntarily participate in this clinical study, abide by the requirements of this clinical study and sign the informed consent.

Exclusion Criteria:

1. Transplanted kidney, severe urinary system deformity, hydronephrosis caused by the compression of tumors of the urinary system and surrounding organs (such as cervical cancer);
2. There are serious diseases in heart, lung, liver and other major organs;
3. Pregnancy;
4. The subject cannot complete the study or comply with the requirements of the study (due to administrative reasons or other reasons).

Ages: 12 Years to 80 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: People aged 12-80 who are scheduled to undergo ureteral stent placement due to urinary calculi, obstruction, etc.; and the estimated time for ureteral stent placement is greater than 2 weeks but less than 1 year.
Sampling Method: Probability Sample
Enrollment: 156 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with ureteral stent encrustation longer than 4mm measured by a ruler | When the patient returns to the hospital to remove the ureteral stent, it may be 2 weeks to 1 year after the operation.
  After indwelling the ureteral stent, ureteral stent encrustation will be formed, which affects the patency of the ureter or causes difficulty in extubation. Our observation outcome is to observe whether the ureteral stent encrustation formed.